CLINICAL TRIAL: NCT01759654
Title: A Trial to Assess the Immunogenicity and Safety of the Trivalent Virosomal Influenza Vaccine, Formulation of 2012-2013, in Non-Elderly Adults and Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLUV12T13A
Record Dates: First submitted 2012-12-17; First posted 2013-01-03 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdimFlu-V (Experimental)
  Interventions: Biological: AdimFlu-V

INTERVENTIONS:
Biological: AdimFlu-V

SUMMARY:
This is an open study of the use of AdimFlu-V (2012-2013 season) vaccine in non-elderly and elderly subjects. All participates will receive one dose of vaccine (0.5 ml) by intramuscular injection into the upper arm. Safety outcomes included immediate reactions at the time of vaccination, solicited local and systemic reactions for 7 days, unsolicited adverse events for 28 days, and serious adverse events. Sera prepared from blood samples will be collected from each subject immediately prior to, and 28 days after vaccination. Anti-hemagglutinin (HA) antibody titers will be determined using the WHO hemagglutination inhibition reference technique. The central laboratory who is responsible for antibody titrations will not be aware of the background of blood samples (e.g., pre- or post-serum), it is also called observer-blinded. All participates will be followed, either by clinical visit or by telephone contact, for 8 weeks after the vaccination for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females and aged no less than 18 years;
2. Willing and able to adhere to visit schedules and all study requirements;
3. Subjects are willing to provide the signed study-specific informed consent.

Exclusion Criteria:

1. Subject or his/her family is employed by the participated hospital;
2. Subjects received influenza vaccine within the previous 6 months;
3. History of hypersensitivity to eggs or hen's protein, polymyxin B, or neomycin, or similar pharmacological effects to study vaccine;
4. Personal or family history of Guillain-Barré Syndrome;
5. An acute febrile illness within 1 week prior to vaccination;
6. Current upper respiratory illness, including the common cold or nasal congestion within 72 hours;
7. Subjects with influenza-like illness as defined by the presence of fever (temperature no less than 38°C) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
8. Female subjects who are pregnant, lactating or likely to become pregnant during the study; women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, intrauterine device (IUD), barrier device or abstinence) throughout the study;
9. Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before study vaccination;
10. Immunodeficiency, or under immunosuppressive treatment;
11. Receipt of live virus vaccine within 1 month prior to study vaccination or expected receipt within 1 month of study vaccination; receipt of any inactivated vaccine within 2 weeks prior to study vaccination or expected receipt within 1 month of study vaccination;
12. Receipt of any blood products, including immunoglobulin in the prior 3 months;
13. Underlying condition in the investigators' opinion may interfere with evaluation of the vaccine;
14. Significant chronic illness for which inactivated influenza vaccine is recommended or commonly used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2012-12-25 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the immune response (i.e. HAI titer) in subjects after administration of influenza vaccine for 2012-2013 season. | Change from baseline for HAI titer at 21 days post immunization
  Serum samples will be obtained prior to vaccination, and 3 weeks post vaccination. Serum samples will be tested for anti-hemagglutinin (HA) antibodies by hemagglutination inhibition (HAI), and assays will be performed at Adimmune Corporation designated central laboratory.

SECONDARY OUTCOMES:
Number of participants reporting reactogenicity events | up to 7 days after vaccination
  Reactogenicity events are pre-specified adverse events systematically recorded on diary cards (a grid of check boxes for each event and each day) during the immediate post-vaccination period by all participants. In general, reactogenicity events will be recorded for 7 days after vaccination. The selection of the events to be collected systematically is based on events expected to occur with wild-type influenza infection including fever (≥38°C), runny nose or nasal congestion, cough, sore throat, muscle aches, headache, vomiting, nausea and malaise. Furthermore, the local (injection site) reactions will also be evaluated that include soreness/pain, swelling, redness, ecchymosis and limitation of arm motion.
Number of participants reporting serious and non-serious adverse events | Up to 8 weeks after vaccination.
  In regard to the long term safety of the study vaccine, the significant and/or serious/non-serious adverse event(s) will be recorded during the 8 weeks follow up after vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan